CLINICAL TRIAL: NCT00352443
Title: Phase I Study Evaluating the Combination of Lapatinib (GW572016; NSC-727989) and Everolimus (RAD001) in Patients With Advanced Solid Tumors
Brief Title: S0528 Lapatinib and Everolimus in Treating Patients With Advanced Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0528; U10CA032102 (NIH); S0528 (Other: SWOG)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia; recurrent adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; unspecified adult solid tumor, protocol specific; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; adult nasal type extranodal NK/T-cell lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, Extranodal NK-T-Cell | interventions — Everolimus; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- everolimus/lapatinib (Experimental): Part 1, dose finding: everolimus and lapatinib at assigned dose daily Part 2, cohort A: Everolimus MTD from Part I: 5 mg PO 1-28 Daily Lapatinib MTD from Part I: 1,250 mg PO Cycle 1, Daily Days 8-28** Subsequent Cycles, Days 1-28 Part 2, cohort B: Lapatinib MTD from Part I: 1,250 mg PO 1-28 Daily Everolimus MTD from Part I: 5 mg PO Cycle 1, Daily Days 8-28** Subsequent Cycles, Days 1-28
  Interventions: Drug: everolimus; Drug: lapatinib ditosylate

INTERVENTIONS:
Drug: everolimus — part 1: dose assigned by ETx online system PO days 1-28 daily part 2: cohort a: 5 mg PO days 1-28 part 2: cohort a: 1250 mg PO days 8-28 (cycle 1) days 1-28 (subsequent cycles)
Drug: lapatinib ditosylate — dose assigned by ETx online system PO days 1-28 daily part 2 cohort a: 1250 mg PO d 8-28 (cycle 1) days 1-28 (subsequent cycles) part 2 cohort b: 120 mg PO days 1-28 daily

SUMMARY:
RATIONALE: Lapatinib and everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Everolimus may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving lapatinib together with everolimus may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib and everolimus in treating patients with advanced solid tumors or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the maximum tolerated dose (MTD) of lapatinib and everolimus in patients with advanced solid tumors or non-Hodgkin's lymphoma. (Part I)
* Investigate the pharmacokinetics of everolimus and lapatinib (when given alone and in combination) at the MTD determined in Part I. (Part II)
* Investigate the effects of everolimus and lapatinib (when given alone and in combination) on serum levels of vascular endothelial growth factor (VEGF), basic fibroblast growth factor (bFGF), matrix metalloproteinase (MMP)-2 and MMP-9, interleukin-6 (IL-6), and tumor necrosis factor alpha (TNF-α). (Part II)

OUTLINE: This is a multicenter, dose-escalation study followed by a randomized study. Initial patients enrolled on the study are treated in part I. After the maximum tolerated dose (MTD) is determined in part I, subsequent patients are enrolled and treated in part II.

* Part I: Patients receive oral everolimus and oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of everolimus and lapatinib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Part II: Patients are randomized to 1 of 2 treatment arms. Everolimus and lapatinib are administered at the MTD determined in part I.

  * Arm I: Patients receive oral everolimus once daily on days 1-28. Patients also receive oral lapatinib once daily on days 8-28 during the first course and on days 1-28 during all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive oral lapatinib once daily on days 1-28. Patients also receive oral everolimus once daily on days 8-28 during the first course and on days 1-28 during all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients in part II undergo blood collection periodically for correlative biomarker and pharmacokinetic studies.

After finishing treatment, patients are followed periodically for 28 days.

PROJECTED ACCRUAL: A total of 48 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor or non-Hodgkin's lymphoma for which no curative options exist
* Measurable or nonmeasurable disease
* Patients with brain metastases who require corticosteroids or anticonvulsants must be on a stable or decreasing dose of corticosteroids and seizure free for 30 days prior to study entry

  * Patients with known brain metastases must have had brain irradiation (whole brain or gamma knife)

    * No untreated (non-irradiated) brain metastases

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Bilirubin normal
* Creatinine normal OR creatinine clearance > 60 mL/min
* Cardiac ejection fraction normal by echocardiogram or MUGA
* Able to swallow enteral medications
* No feeding tubes
* No intractable nausea or vomiting
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication
* No current active hepatic or biliary disease with the exception of Gilbert's syndrome or asymptomatic gallstones
* No malabsorption syndrome
* No requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or everolimus, including other quinazoline compounds, such as gefitinib and erlotinib, or other rapamycins, such as sirolimus and temsirolimus
* No known HIV positivity
* No concurrent uncontrolled illness, including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction or cerebrovascular accident within the past 3 months
  * Uncontrolled diarrhea
  * Psychiatric illness or social situation that would preclude compliance with study requirements
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to undergo pharmacokinetic (PK) sampling and blood collection for PK and correlative studies (for patients enrolled in part II)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior lapatinib or everolimus
* No prior surgical procedures affecting absorption
* More than 14 days since prior major surgery, chemotherapy (42 days for nitrosoureas or mitomycin C), or radiotherapy
* More than 28 days since prior investigational agents
* At least 7 days since prior and no concurrent CYP3A4 inhibitors
* At least 14 days since prior and no concurrent CYP3A4 inducers
* At least 14 days since prior and no concurrent herbal or dietary supplements
* No concurrent chemotherapy, hormone therapy, radiotherapy, immunotherapy, live vaccines or any other anticancer therapy

  * Concurrent luteinizing hormone-releasing hormone agonists allowed
  * Concurrent bisphosphonates or epoetin alfa or its analogue allowed
* No concurrent gastric H2 blockers (e.g., cimetidine, ranitidine, nizatidine, famotidine) or proton pump inhibitors (e.g., omeprazole, esomeprazole, rabeprazole, pantoprazole, or lansoprazole)

  * Antacids allowed provided they are not administered within 1 hour before and after lapatinib
* No concurrent glucocorticoids or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of lapatinib and everolimus (Part I) | 1 month

SECONDARY OUTCOMES:
Pharmacokinetics (Part II) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute; Patricia M. LoRusso, DO, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (6):
- United States (6):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Hoban CJ, Hoering A, Synold TW, et al.: Phase I evaluation of lapatinib and everolimus in patients with advanced malignancies: Southwest Oncology Group trial S0528. [Abstract] J Clin Oncol 27 (Suppl 15): A-3553, 2009.
- [Derived] Gadgeel SM, Lew DL, Synold TW, LoRusso P, Chung V, Christensen SD, Smith DC, Kingsbury L, Hoering A, Kurzrock R. Phase I study evaluating the combination of lapatinib (a Her2/Neu and EGFR inhibitor) and everolimus (an mTOR inhibitor) in patients with advanced cancers: South West Oncology Group (SWOG) Study S0528. Cancer Chemother Pharmacol. 2013 Nov;72(5):1089-96. doi: 10.1007/s00280-013-2297-4. Epub 2013 Sep 22. PMID 24057042